CLINICAL TRIAL: NCT07011017
Title: Sexual Health of Sub-Saharan African Migrant Women Recently Diagnosed With HIV in Île-de-France: Missed Opportunities for Prevention
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0078.1_SMIT_FASVIH
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections; Sexual Health; Migrants; Women's Health; Health Services Accessibility; Sub-Saharan Africa; Risk-Taking; Vulnerable Populations
MeSH Terms: conditions — HIV Infections; Risk-Taking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
This study looks at the sexual health of women from Sub-Saharan Africa who recently found out they have HIV after arriving in Île-de-France. It aims to understand their risk factors and identify missed chances for HIV testing and prevention. The goal is to improve care and support for these women by learning more about their experiences and the challenges they face.

ELIGIBILITY:
Inclusion Criteria:

* Sub-Saharan African migrant women recently diagnosed with HIV (from 2021 onward)
* HIV diagnosis made on French territory
* Aged 18 years or older

Exclusion Criteria:

* Inability to inform the patient about the study due to a language barrier or other obstacle
* HIV diagnosis made before 2021
* HIV diagnosis made in the country of origin
* Under 18 years of age

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study population will consist of Sub-Saharan African migrant women living in Île-de-France who were newly diagnosed with HIV on French territory from 2021 onward. Participants will be selected from two infectious disease departments: the SMIT at the Centre Hospitalier Sud Francilien (CHSF) and the SMIT at the hospital in Melun. Eligible participants must be at least 18 years old and meet the inclusion criteria. This population is particularly vulnerable due to social, economic, and structural barriers that may limit access to sexual health services and HIV prevention.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Description of sexual health characteristics (e.g., history of sexually transmitted infections, contraceptive use, number and type of sexual partners, presence of transactional sex, and access to sexual health services) in Sub-Saharan African migrant wom | enrollment - 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France